CLINICAL TRIAL: NCT05880251
Title: Operant Conditioning of Sensory Evoked Potentials to Reduce Phantom Limb Pain
Brief Title: Operant Conditioning of Sensory Brain Responses to Reduce Phantom Limb Pain in People With Limb Amputation
Acronym: OCS-PLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F4410-P; 1I21RX004410-01A1 (NIH)
Record Dates: First submitted 2023-05-09; First posted 2023-05-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Phantom Limb Pain After Amputation; Lower Limb Amputation; Upper Limb Amputation; Phantom Pain; Chronic Pain
Keywords: Phantom limb pain; Amputation; Operant Conditioning; Brain-Computer Interface; Electroencephalography; Tactile sense; Instrumental learning; Event Related Potentials
MeSH Terms: conditions — Phantom Limb; Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to 2 groups, one group receiving the operant conditioning feedback with peripheral stimulation (Intervention group) and the other receiving only peripheral stimulation with no operant conditioning feedback (Control group).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The pre and post clinical assessment will be performed by a blinded evaluator.
  * The participant will not be told about group assignment till the end of the last follow-up session and assessment
  * Investigators will keep blinded to the baseline clinical measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Intervention group receives peripheral stimulation with realtime operant conditioning feedback training.
  Interventions: Behavioral: Operant Conditioning with Peripheral Stimulation
- Control Group (Experimental): Control group receives peripheral stimulation but without operant conditioning feedback.
  Interventions: Behavioral: Control Group with Peripheral Stimulation Only

INTERVENTIONS:
Behavioral: Operant Conditioning with Peripheral Stimulation — This is a training intervention to strengthen the weakened sensorimotor responses and reduce pain, after a limb amputation. Non-painful peripheral stimulation will be applied to elicit a response.
  Arms: Intervention Group
Behavioral: Control Group with Peripheral Stimulation Only — This is a control intervention in which the non-painful peripheral stimulation will be applied, same as the operant conditioning group, but no training feedback will be provided.
  Arms: Control Group

SUMMARY:
The study will investigate the application of a non-pharmacological operant conditioning approach to reduce phantom limb pain (PLP). PLP afflicts 60-90% people who have lost a limb. It can last for years and lead to drug dependence, job loss, and poor quality of life. Current non-pharmacological interventions are encouraging but limited, and their efficacy remains unclear. Limb amputation is known to lead to abnormal sensorimotor reorganization in the brain. Multiple studies have shown that PLP severity is correlated with the extent of this reorganization. The current study will train participants via realtime feedback of brain responses to promote more normal sensorimotor response, with the goal to reduce phantom limb pain.

DETAILED DESCRIPTION:
The study will be recruiting people who have had a limb amputation (traumatic or atraumatic) and are experiencing chronic phantom limb pain (PLP). Participants will be asked to be seated during the study session. Non-painful peripheral stimulation will be applied to elicit an evoked response (from either muscle or brain). Electrodes will be placed on the muscles and or scalp to record these electrical brain responses during the study session. Visual feedback based on the response will be provided in pseudo realtime. The study will involve three 1-hour sessions per week for 8-9 weeks, followed by 2 follow-up sessions at 3 and 6 months after the last session. Assessments of pain intensity and quality, and neurophysiological sensorimotor response, will be performed before the first session, after the last session, and at follow-up sessions. Additional electroencephalography (EEG) based assessments will also be performed as exploratory measures, to assess inter- and intra- hemispheric functional connectivity and sensorimotor responses associated with amputation and operant conditioning training.

ELIGIBILITY:
Inclusion Criteria:

* An upper (or lower limb) amputation more than 6 months ago, that has produced a moderate to severe hand/arm (or foot/leg) phantom limb pain,
* Male or female age 18 years or older,
* Medical clearance to participate,
* Reasonable expectation that ongoing medications, if any, will be maintained without change for at least 4 months from the start of the study,
* Able to provide informed consent and to understand the study instructions,
* Able to participate in the specific study procedures.

Exclusion Criteria:

* Presence of other medically unstable and/or infectious condition (e.g., uncontrolled diabetes with recent weight loss, diabetic coma, frequent insulin reactions),
* A cardiac condition (e.g., history of myocardial infarction or congestive heart failure),
* Cognitive and/or attention difficulties affecting participant's ability to follow study directions,
* Known skin disorders or damaged skin at the anticipated at the scalp for EEG recording (e.g., unhealed wounds, broken skin).
* Metal implants above the chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Change in Pain as Measured by the Short form-McGill Pain Questionnaire (SF-MPQ) | Baseline, end of training (session 20) i.e. approximately 10 weeks from baseline, follow-up at 3-months after training ends, follow-up at 6-months after training ends
  The Sf-MPQ assesses the pain quality in the sensory (11 items) and affective (4 items) dimensions. Each item is rated on an intensity scale of 0 (none) to 3 (severe). Total score is obtained by summing the scores for all items and the range is 0 (no pain) to 45 (severe pain).
Change in Evoked Potential (EP) Amplitude and threshhold | Baseline, end of training (session 20) i.e. approximately 10 weeks from baseline, follow-up at 3-months after training ends, follow-up at 6-months after training ends
  The evoked response to tactile stimuli will be captured in one of two ways 1) EMG and Reflex evoke responses from cutaneous nerve on the residual Limb and 2) With 64 channel non-invasive scalp electroencephalography (EEG) electrodes placed on the scalp. SSEP will be assessed at the sensorimotor cortex contralateral to the amputated limb. An increase in amplitude will indicate improvement in the sensorimotor response and tolerance.
Change in Somatosensory Evoked Potential (SSEP) Latency as Measured by a Tactile Event Related Potential Test | Baseline, end of training (session 20) i.e. approximately 10 weeks from baseline, follow-up at 3-months after training ends, follow-up at 6-months after training ends
  The evoked response to tactile stimuli will be captured with 64 channel non-invasive scalp electroencephalography (EEG) electrodes placed on the scalp. SSEP will be assessed at the sensorimotor cortex contralateral to the amputated limb. A reduction in latency will indicate improvement in the sensorimotor cortical response.

SECONDARY OUTCOMES:
Change in Impact of Pain on Quality of Life as Measured by the West Haven-Yale Multidimensional Pain Inventory (WHYMPI) | Baseline, end of training (session 20) i.e. approximately 10 weeks from baseline, follow-up at 3-months after training ends, follow-up at 6-months after training ends
  This is a 52-item inventory with 12 subscales over 3 domains. Each item is scored on a 0-6 scale. Scores for each subscale are obtained by taking the mean of the scores of all items in that subscale. Higher scores indicate more severity in that subscale.
  Part I includes five scales designed to measure important dimensions of the chronic pain experience; Part II assesses patients' perceptions of the degree to which spouses or significant others display Solicitous, Distracting or Negative responses to their pain behaviors and complaints. Part III assesses patients' report of the frequency with which they engage in four categories of common everyday activities; Household Chores, Outdoor Work, Activities Away from Home, and Social Activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi A Brangaccio, PT, Principal Investigator — Albany VA Medical Center Samuel S. Stratton, Albany, NY
Locations (1):
- Albany VA Medical Center Samuel S. Stratton, Albany, NY, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson AK, Wolpaw JR. Operant conditioning of spinal reflexes: from basic science to clinical therapy. Front Integr Neurosci. 2014 Mar 18;8:25. doi: 10.3389/fnint.2014.00025. eCollection 2014. PMID 24672441

DOCUMENTS (1):
  • Informed Consent Form (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT05880251/ICF_000.pdf